CLINICAL TRIAL: NCT00213122
Title: Effects of Miglitol on Daily Plasma Glucose in type2 Diabetes Treated With Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MG1007
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-09-28 (Estimated); Status verified 2006-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: alpha-glucosidase inhibitor,Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — miglitol

INTERVENTIONS:
Drug: miglitol

SUMMARY:
In this study, the effect of miglitol on daily plasma glucose will be evaluated in type 2 diabetic patients treated with insulin.

ELIGIBILITY:
Inclusion Criteria:

* type2 diabetes
* postprandial plasma glucose levels ≧180mg/dl

Exclusion Criteria:

* type1 diabetes
* AST(GOT) or ALT(GPT) ≧100IU/l
* creatinine ≧2.0mg/dl

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Promotiom Group, Study Director — Sanwa Kagaku Kenkyusho Co., Ltd.
Locations (1):
- Ibaraki, Japan